CLINICAL TRIAL: NCT01946399
Title: Dexamethasone Intravitreal Implant for Retinal Vein Occlusion Associated Macular Edema After Treatment Failure With Anti-VEGF Medications
Brief Title: Ozurdex Implant for Macular Edema After Treatment Failure With Anti-VEGF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment not met
Sponsor: Retina Research Institute, LLC (Other)
Collaborators: Retina-Vitreous Associates Medical Group (Other); West Coast Retina Medical Group, Inc. (Other)
Responsible Party: Principal Investigator, Rhonda Weeks, Gaurav K. Shah, MD, Retina Research Institute, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ozurdex RVO 2013
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Retinal Vein Occlusion (RVO); Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ozurdex implant (Other): Intravitreal injection of Ozurdex implant
  Interventions: Drug: Ozurdex implant

INTERVENTIONS:
Drug: Ozurdex implant — Intravitreal injection of Dexamethasone implant
  Other Names: Dexamethasone implant

SUMMARY:
To determine if Ozurdex implant can offer an effective treatment for macular edema associated with retinal vein occlusion when treatment with intravitreal Avastin, Lucentis, or Eylea have not demonstrated a significant response.

DETAILED DESCRIPTION:
To determine whether Ozurdex implant can offer an efficacious alternative for treatment of macular edema in the setting of retinal vein occlusion when treatment with intravitreal bevacizumab (Avastin),ranibizumab (Lucentis), and/or aflibercept (Eylea) have not demonstrated significant response.

ELIGIBILITY:
Inclusion Criteria:

All patients with Retinal Vein Occlusion (RVO) with available initial imaging and documented treatment failure with bevacizumab, ranibizumab, or aflibercept. Treatment failure is defined as lack of anatomic improvement (persistent intraretinal cystic changes/macular edema with central subfield thickness greater than 250 microns on time-domain OCT or greater than 275 microns on spectral domain OCT) with lack of visual improvement (less than 2 lines of visual gain by Snellen acuity), despite 3 to 6 intravitreal anti-VEGF treatments over the preceding 6 months.

Exclusion Criteria:

* Co-existing or pre-existing macular degeneration, diabetic macular edema, or other confounding disease processes
* Interval surgical intervention, such as cataract surgery, that may confound visual outcomes.
* Pregnancy
* Coexisting conditions that would represent relative or absolute contraindications usage of ozurdex implant, including:
* Ocular or periocular infections (including viral disease of the cornea and conjunctiva such as active epithelial herpes simplex keratitis, vaccinia, varicella, mycobacterial infection, and fungal diseases)
* Advanced glaucoma
* Aphakic eyes with rupture or missing posterior lens capsule
* Eyes with anterior chamber intraocular lens and missing posterior lens capsule
* Patients with known hypersensitivity to components of this product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Improvement in best-corrected Snellen visual acuity following initiation of Ozurdex therapy | 6 Months

SECONDARY OUTCOMES:
Anatomic/angiographic improvement in macular edema as evaluated by OCT and fluorescein angiography | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav K Shah, MD, Principal Investigator — Retina Research Institute
Locations (1):
- The Retina Institute, St Louis, Missouri, United States